CLINICAL TRIAL: NCT01288170
Title: Pharmacokinetic Bioequivalence Study of Nebcinal® 150mg/3ml Administered by Aeroneb® Idehaler® Versus Tobi® 300mg/5ml Administered by Pari LC Plus®
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Erempharma (Industry)
Collaborators: Hospices Civils de Lyon (Other); University of Lyon (Other)
Responsible Party: Jean Pierre Salin, EREMPHARMA
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RM/NEB-02/09
Record Dates: First submitted 2011-02-01; First posted 2011-02-02 (Estimated); Last update posted 2011-02-02 (Estimated); Status verified 2011-02

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis, bioequivalence, pharmacokinetic, sputum, plasma
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nebcinal Tobi (Other): crossover design
  Interventions: Drug: Nebcinal Tobi
- Tobi Nebcinal (Other): crossover design
  Interventions: Drug: Tobi Nebcinal

INTERVENTIONS:
Drug: Nebcinal Tobi
  Arms: Nebcinal Tobi
Drug: Tobi Nebcinal
  Arms: Tobi Nebcinal

SUMMARY:
Cystic fibrosis (CF) is a genetic disease characterized by mutations in CFTR (Cystic Fibrosis Transmembrane conductance Regulator) gene. Mortality and morbidity are mostly related to the respiratory affection which appears early in neonates.

The constant improvement in symptomatic treatments and care strategies allowed CF patients' life expectancy to be increased over the last decades.

Vital prognostic is related to bronchopulmonary infections. 39% of CF patients under 18 years old and 70% of adult CF patients are chronically infected by Pseudomonas aeruginosa.

Elevated concentrations of tobramycin in broncho secretions, about 1000 times the MIC, is obtained by inhaled administration of tobramycin and is active against in vitro resistant Pseudomonas aeruginosa.

Study hypotheses :

Regarding literature data and in vitro studies, the administration of Nebcinal® 150mg/3ml administered twice a day by Aeroneb® Idehaler® pocket® would deliver the same quantity of antibiotic in lung and plasma as Tobi® 300mg/5ml administered twice a day by Pari® LC Plus® in children and adult patients with CF.

Primary objective :

To compare plasma concentrations after inhalation of Nebcinal® 150mg/3ml administered by Aeroneb® Idehaler pocket® and Tobi® 300 mg/5ml administered by Pari LC Plus®

ELIGIBILITY:
Inclusion Criteria:

* Adults and children aged 6 years old and more
* Male or female
* Patients with cystic fibrosis (positive sudoral test, Cl > 60 mmol/L)
* Followed in a CRCM (CF care centre)
* FEV1 ≥40%
* Informed consent collected from adults or parents or legal guardians and children.
* Affiliation to the National Health Insurance program (Sécurité sociale).

Exclusion Criteria:

* - renal insufficiency defined by a creatinine clearance level superior to 2 mg/dl
* recent pneumothorax, emphysema, punction or recent pleural biopsy, recent haemoptysis superior to 60 ml within 30 days prior to randomization
* Acute pulmonary exacerbation pathology, according to conference of consensus (2002), evaluated by :

Cough increase, Sputum increase, Decrease in tolerance to effort, Loss of weight, lack of appetite, Deterioration of respiratory function,

- Medical history of intolerance, toxicity or allergy to tobramycine, hypersensitivity to aminoside

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2010-02; Primary Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
plasma Area under the curve from 0 to 8 hours of tobramycine after administration of the drug

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre de ressources et de compétences pour la mucovisidose, enfants, Bron
  - Centre de ressources et de compétences pour la mucovisidose, adultes, Pierre-Bénite